CLINICAL TRIAL: NCT07338786
Title: A Single-Center, Open-Label, Single-Arm, Phase I Clinical Trial to Evaluate the Safety of a Lyophilized Human Rabies Vaccine (Human Diploid Cell) Administered in Different Immunization Schedules.
Brief Title: A Phase I Clinical Trial to Evaluate the Safety of Different Immunization Schedules of a Lyophilized Human Rabies Vaccine (Human Diploid Cell)
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Changchun BCHT Biotechnology Co. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B1901-F20230313-1
Record Dates: First submitted 2026-01-04; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: RabiesPrevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lyophilized Human Rabies Vaccine (Human Diploid Cell) (Experimental)
  Interventions: Drug: Lyophilized Human Rabies Vaccine (Human Diploid Cell)

INTERVENTIONS:
Drug: Lyophilized Human Rabies Vaccine (Human Diploid Cell) — Each human dose is 0.5 ml.

SUMMARY:
This clinical trial employed a single-center, open-label, single-arm design. A total of 80 participants aged 10 to 60 years were enrolled and divided into two age groups: 40 in the 18-60 years cohort and 40 in the 10-17 years cohort. All participants received the lyophilized human rabies vaccine (human diploid cell)

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 10 to 60 years;
* Informed consent can be obtained from the participant and/or their guardian;
* The participant and/or guardian are able to comply with the requirements of the clinical trial protocol.

Exclusion Criteria:

* Axillary temperature>37.0°C on the day of vaccination
* History of rabies vaccination or use of rabies virus passive immunization preparations
* History of dog or other mammalian bites or scratches (with skin laceration) within 1 year prior to the first vaccination
* Abnormalities in laboratory tests such as complete blood count (CBC), blood biochemistry, and urinalysis before the first vaccination are clinically significant and cannot be excluded based on the investigator's comprehensive assessment.
* Suffering from acute illness or acute exacerbation of chronic disease within 3 days prior to the first vaccination
* Urinary pregnancy test results were positive in female participants of childbearing age, or they were in the lactation period, or female participants of childbearing age, male participants, or their partners had fertility plans during the trial period.
* History of severe allergic reactions requiring medical intervention or severe adverse reactions to vaccines (e.g., severe urticaria, anaphylactic shock, allergic laryngeal edema, Henoch-Schönlein purpura, localized allergic necrotic reaction (Arthus reaction), angioedema, etc.), or allergy to any component of the trial vaccine, such as human serum albumin, dextran 40, sucrose, glycine, disodium hydrogen phosphate, or potassium dihydrogen phosphate.
* Known or suspected malignancy, autoimmune disease, immunodeficiency, or immunosuppression (e.g., human immunodeficiency virus (HIV) infection, organ transplantation, systemic lupus erythematosus (SLE), rheumatoid arthritis, etc.)
* Within 6 months prior to the first dose or with a planned long-term use of immunosuppressants and/or immunomodulators (e.g., systemic glucocorticoids, continuous use of targeted immunomodulators for more than 14 days), cytotoxic therapy, etc.
* Patients with congenital malformations or developmental disorders affecting organ function, uncontrolled hypertension (limited to 18-60 years of age) [maintained with medication at systolic blood pressure ≥140 mmHg and/or diastolic blood pressure ≥90 mmHg], severe hepatic or renal diseases (critical cases, e.g., with concomitant diabetes), etc.
* Contraindications to intramuscular injection, such as local infection or skin lesions at the injection site, severe thrombocytopenia, coagulation dysfunction, or a history of coagulation disorders
* History or family history of psychiatric and neurological disorders such as convulsions, epilepsy, encephalopathy, and psychosis
* Individuals who have received or plan to use blood products or immunoglobulin products during the trial period within the past 3 months
* Received other investigational drugs within 1 month prior to trial vaccine administration or was participating in other clinical trials
* Received a live attenuated vaccine within 14 days prior to enrollment, or a subunit or inactivated vaccine within 7 days prior to enrollment

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-13 (Actual); Primary Completion 2026-01-04 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Safety Endpoints | within 30 Days After last Vaccination
  Incidence of Adverse Events within 30 Days After last Vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu CDC, Xuzhou, Jiangsu, China